CLINICAL TRIAL: NCT00654407
Title: An Open Label, Randomized, Multi-Center, Phase IIIB, Parallel Group Switching Study to Compare the Efficacy and Safety of Lipid Lowering Agents Atorvastatin and Simvastatin With Rosuvastatin in High Risk Subjects With Type IIa and IIb Hypercholesterolemia.
Brief Title: Mercury II - Compare the Efficacy and Safety of Lipid Lowering Agents Atorvastatin and Simvastatin With Rosuvastatin in High Risk Subjects With Type IIa and IIb Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4522IL/0068; D3560C00068
Record Dates: First submitted 2008-04-03; First posted 2008-04-08 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia
Keywords: Cholesterol; hypercholesterolemia; Coronary Heart disease; low density lipoproteins; Rosuvastatin; Atorvastatin; simvastatin
MeSH Terms: conditions — Hypercholesterolemia; Coronary Disease | interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (Active Comparator): Atorvastatin
  Interventions: Drug: Atorvastatin
- 3 (Active Comparator): Simvastatin
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Drug: Atorvastatin
  Other Names: Lipitor
  Arms: 2
Drug: Simvastatin
  Other Names: Zocor
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether treatment with rosuvastatin following atorvastatin or simvastatin treatment will improve health outcomes for patients at high risk of Coronary heart disease compared to atorvastatin and simvastatin alone.

ELIGIBILITY:
Inclusion Criteria:

* Discontinuation of all cholesterol lowing drugs, including dietary supplements.
* Documented history of, or high risk of coronary heart disease or other established atherosclerotic disease.

Exclusion Criteria:

* The use of lipid lowering drugs or dietary supplements after Visit 1.
* Active arterial disease eg Unstable angina, or recent arterial surgery
* Uncontrolled hypertension, hypothyroidism, alcohol or drug abuse.
* Abnormal laboratory parameters as defined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4875 (Estimated)
Dates: Start 2001-11; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Low density Lipoprotein cholesterol level - reaching internationally recognised LDL cholesterol goal levels. | 16 weeks

SECONDARY OUTCOMES:
Percentage change in other cholesterol & triglyceride measures | 16 weeks
Safety evaluation | 8 & 16 weeks
To compare the efficacy of rosuvastatin with atorvastatin and simvastatin

CONTACTS AND LOCATIONS:
Overall Officials: Joel Raichlen, Study Director — AstraZeneca; Russell Esterline, Study Director — AstraZeneca

REFERENCES:
- [Derived] Ballantyne CM, Raichlen JS, Cain VA. Statin therapy alters the relationship between apolipoprotein B and low-density lipoprotein cholesterol and non-high-density lipoprotein cholesterol targets in high-risk patients: the MERCURY II (Measuring Effective Reductions in Cholesterol Using Rosuvastatin) trial. J Am Coll Cardiol. 2008 Aug 19;52(8):626-32. doi: 10.1016/j.jacc.2008.04.052. PMID 18702965